CLINICAL TRIAL: NCT01038713
Title: A Prospective Randomized Trial of Plastic vs. Covered Metal vs. Uncovered Metal Biliary Stents for the Management of Malignant Biliary Obstruction
Brief Title: Plastic vs. Covered Metal vs. Uncovered Metal Biliary Stents for the Management of Malignant Biliary Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-01
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Resectable; plastic stent (Experimental): Patients determined to have surgically resectable malignancy presenting with malignant biliary obstruction randomized to receive a plastic biliary stent to relieve their biliary obstruction.
  Interventions: Device: Biliary stent placement
- Resectable; uncovered metal stent (Experimental): Patients determined to have surgically resectable malignancy presenting with malignant biliary obstruction randomized to receive an uncovered metal biliary stent to relieve their biliary obstruction.
  Interventions: Device: Biliary stent placement
- Resectable; fully covered metal stent (Experimental): Patients determined to have surgically resectable malignancy presenting with malignant biliary obstruction randomized to receive a fully-covered metal biliary stent to relieve their biliary obstruction.
  Interventions: Device: Biliary stent placement
- Unresectable; uncovered metal stent (Experimental): Patients determined to have surgically non-resectable malignancy presenting with malignant biliary obstruction randomized to receive an uncovered metal biliary stent to relieve their biliary obstruction.
  Interventions: Device: Biliary stent placement
- Unresectable; fully covered metal stent (Experimental): Patients determined to have surgically non-resectable malignancy presenting with malignant biliary obstruction randomized to receive a fully-covered metal biliary stent to relieve their biliary obstruction.
  Interventions: Device: Biliary stent placement

INTERVENTIONS:
Device: Biliary stent placement — Patient's with a malignant biliary obstruction will undergo placement of a biliary stent via ERCP.

SUMMARY:
This is a single center, randomized, unblinded study to compare the rate of occlusion of plastic, uncovered metal, or fully covered metal biliary stents in patient's with surgically resectable disease or those undergoing neoadjuvant chemoradiotherapy. We will also compare occlusion rates between uncovered metal and fully covered metal biliary stents in those patients determined to have surgically unresectable disease.

DETAILED DESCRIPTION:
Malignant biliary obstruction can result from extrinsic processes, such as proximal pancreatic ductal adenocarcinoma or metastatic lesions, or from intrinsic lesions such as cholangiocarcinoma. Malignant biliary obstruction is typically treated endoscopically with placement of either plastic (polyethylene) or metal biliary stents. Metal stents have a wider diameter than plastic stents, and have been shown to have higher patency rates, but are also 15-40 times the cost of plastic stents. Metal stents with a polymer coating have been developed to prevent tumor ingrowth into the stent, which can lead to stent occlusion. Cost analysis has demonstrated an advantage to the use of metal stents in patients with unresectable disease, or who may achieve operable status following neoadjuvant chemotherapy, while either plastic stents or metal stents are used when patients are deemed to have a surgically resectable lesion. Patient's determined to have resectable, or borderline resectable malignancy (those who may achieve resectability status following neoadjuvant chemotherapy) will receive either plastic, uncovered metal, or covered metal stents in a randomized fashion, while patients determined to have surgically unresectable malignancy will randomly receive either covered or uncovered metal biliary stents. The primary aim of this study is to prospectively evaluate stent occlusion rates in patients presenting with malignant biliary obstruction. Secondary aims of the study will include a cost analysis of each stent type, rate of hospital admission following stent placement, days off of chemotherapy due to procedural complication, and rate of acute cholecystitis associated with stent placement.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female older than 18
2. Capable of providing written informed consent
3. Presenting with malignant biliary obstruction requiring biliary drainage either from proximal pancreatic malignancy, metastatic disease, or intrinsic biliary malignancy. The patient must have an established diagnosis of underlying malignancy, and surgical resectability status established, prior to enrollment in this study.

Exclusion Criteria

1. Inability to undergo conscious sedation or monitored anesthesia
2. Prior pancreatico-biliary surgery
3. Evidence of acute cholecystitis at time of endoscopic procedure
4. Intraluminal filling defect requiring endoscopic removal prior to stent placement
5. Inability to provide written informed consent
6. Malignancy not verified prior to stent placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Gardner, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Gardner TB, Spangler CC, Byanova KL, Ripple GH, Rockacy MJ, Levenick JM, Smith KD, Colacchio TA, Barth RJ, Zaki BI, Tsapakos MJ, Gordon SR. Cost-effectiveness and clinical efficacy of biliary stents in patients undergoing neoadjuvant therapy for pancreatic adenocarcinoma in a randomized controlled trial. Gastrointest Endosc. 2016 Sep;84(3):460-6. doi: 10.1016/j.gie.2016.02.047. Epub 2016 Mar 10. PMID 26972022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol initially was designed to measure five groups - we elected not to study patients with unresectable disease and thus only patients with presumed resectable disease are included
Pre-assignment Details: 94 patients recruited for the study. 63 were randomized into three arms
Period: Overall Study
Arm/Group | Resectable; Plastic Stent | Resectable; Uncovered Metal Stent | Resectable; Fully Covered Metal Stent
Started | 26 | 20 | 17
Completed | 21 | 17 | 16
Not Completed | 5 | 3 | 1
Not completed — Patient to hospice | 1 | 1 | 1
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Neuroendocrine Tumor | 0 | 1 | 0
Not completed — died from PEP | 0 | 1 | 0
Not completed — Autoimmune Pancreatitis | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resectable; Plastic Stent | Resectable; Uncovered Metal Stent | Resectable; Fully Covered Metal Stent | Total
Number analyzed (Participants) | 21 | 17 | 16 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (9.67) | 64.8 (8.47) | 67.2 (11.4) | 65.9 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 7 | 23
  Male | 11 | 11 | 9 | 31
Region of Enrollment [Number; unit: participants]
  United States | 21 | 17 | 16 | 54

OUTCOME MEASURES:

1. Primary Outcome: Assess the Occlusion Rates, Attempted Surgical Resection or Death of Plastic, Covered, and Uncovered Biliary Stents in Patients Presenting With Malignant Biliary Obstruction.
Description: Number of participants who developed stent occlusion, attempted surgical resection or death following stent placement
Time Frame: Time of stent occlusion, attempted surgical resection or patient death to 300 days
Measure: Number; unit: participants
Arm/Group | Resectable; Plastic Stent | Resectable; Uncovered Metal Stent | Resectable; Fully Covered Metal Stent
Number analyzed (Participants) | 21 | 17 | 16
participants
  Stent Occlusion | 11 | 6 | 4
  Attempted Surgical Resection | 4 | 6 | 8
  Death | 6 | 5 | 4
Statistical Analysis 1: Comparison: Resectable; Plastic Stent vs Resectable; Uncovered Metal Stent vs Resectable; Fully Covered Metal Stent; Test type: Superiority or Other; p = 0.22, Chi-squared — Analysis comparing the number of patients who had stent occlusion; 3 x 2 contingency table comparing all three groups
Statistical Analysis 2: Comparison: Resectable; Plastic Stent vs Resectable; Uncovered Metal Stent vs Resectable; Fully Covered Metal Stent; Analysis comparing the rate of attempted surgical resection; Test type: Superiority or Other; p = 0.14, Chi-squared; 3 x 2 contingency table comparing all three groups
Statistical Analysis 3: Comparison: Resectable; Plastic Stent vs Resectable; Uncovered Metal Stent vs Resectable; Fully Covered Metal Stent; Analysis comparing the rate of death between groups; Test type: Superiority or Other; p = 0.96, Chi-squared; 3 x 2 contingency table comparing all three groups

2. Secondary Outcome: Total Cost Associated With the Placement of Biliary Stents Including the Cost of the Device as Well as the Secondary Costs of Device Placement.
Time Frame: Costs measured up to 500 days
Measure: Number; unit: United States Dollars
Arm/Group | Resectable; Plastic Stent | Resectable; Uncovered Metal Stent | Resectable; Fully Covered Metal Stent
Number analyzed (Participants) | 21 | 17 | 16
United States Dollars | 39,955 | 41,476 | 41,112
Statistical Analysis 1: Comparison: Resectable; Plastic Stent vs Resectable; Uncovered Metal Stent vs Resectable; Fully Covered Metal Stent; Test type: Superiority or Other; p = 1.00, ANOVA

3. Secondary Outcome: Determine the Days of Hospitalization Following Stent Placement
Description: Number of total days of hospitalization for all patients in each group
Time Frame: From stent placement up to 500 days post stent
Measure: Number; unit: Days
Arm/Group | Resectable; Plastic Stent | Resectable; Uncovered Metal Stent | Resectable; Fully Covered Metal Stent
Number analyzed (Participants) | 21 | 17 | 16
Days | 0 | 14 | 15

4. Secondary Outcome: Assess Days Neoadjuvant Therapy Was Delayed Due to Complications Associated With the Stents
Description: Total number of days in which neoadjuvant therapy was delayed due to stent related issues
Time Frame: Time from stent placement to 500 days
Measure: Number; unit: Days
Arm/Group | Resectable; Plastic Stent | Resectable; Uncovered Metal Stent | Resectable; Fully Covered Metal Stent
Number analyzed (Participants) | 21 | 17 | 16
Days | 73 | 50 | 3

5. Secondary Outcome: Assess Rate of Acute Cholecystitis Associated With Each Type of Stent
Time Frame: time from stent placement to 500 days
Measure: Number; unit: Participants
Arm/Group | Resectable; Plastic Stent | Resectable; Uncovered Metal Stent | Resectable; Fully Covered Metal Stent
Number analyzed (Participants) | 21 | 17 | 16
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Time from stent placement to 500 days
Arm/Group | Resectable; Plastic Stent | Resectable; Uncovered Metal Stent | Resectable; Fully Covered Metal Stent
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/21 | 3/17 | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Resectable; Plastic Stent (N=21) | Resectable; Uncovered Metal Stent (N=17) | Resectable; Fully Covered Metal Stent (N=16)
Post-ERCP Pancreatitis (Gastrointestinal disorders) | 0 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes